CLINICAL TRIAL: NCT07033247
Title: The Effect of Different Sodium Hypochlorite Concentrations and Activation Techniques on Postoperative Pain in Permanent Molars With Chronic Apical Periodontitis: A Randomized Controlled Trial
Brief Title: The Effect of Different Sodium Hypochlorite Concentrations and Activation Techniques on Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Kübra Gürler, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 08.11.2024/149
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Chronic Apical Periodontitis
Keywords: Sodium hypochlorite; Chronic apical periodontitis; Postoperative pain; Irrigation activation; Passive ultrasonic irrigation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 2.5% NaOCl - Neddle Irrigation (No Intervention): Irrigation was performed with a 30 G side-vented needle using 2.5% sodium hypochlorite (NaOCl). A total of 11 mL NaOCl was used: 2 mL after coronal preparation, 2 mL after middle third, 2 mL after apical third preparation, and 5 mL as final irrigation. Canals were then flushed with 2 mL saline and 2 mL 17% Ethylenediaminetetraacetic Acid (EDTA).
- 2.5% NaOCl - EDDY Activation (Experimental): Following 2 mL irrigation with 2.5% NaOCl, canals were activated using the EDDY sonic system (25/04 polyamide tip, 6000 Hz) 2 mm short of working length for 20 seconds, repeated 3 times. Between activations, 1 mL NaOCl was used. Total 11 mL NaOCl was delivered. Final irrigation was performed with 2 mL saline and 2 mL 17% EDTA.
  Interventions: Device: EDDY Sonic Activation System
- 2.5% NaOCl - Passive Ultrasonic Irrigation (Experimental): Canals were irrigated with 2 mL 2.5% NaOCl and activated using a passive ultrasonic tip without contact with dentin walls, 2 mm short of working length for 20 seconds, repeated 3 times. Each cycle was followed by 1 mL NaOCl. Final irrigation included 2 mL saline and 2 mL 17% EDTA.
  Interventions: Device: Passive Ultrasonic Irrigation (PUI)
- 5.25% NaOCl - Needle Irrigation (No Intervention): Irrigation was performed with a 30 G side-vented needle using 5.25% sodium hypochlorite. A total of 11 mL NaOCl was used as in the other groups. Final irrigation included 2 mL saline and 2 mL 17% EDTA.
- 5.25% NaOCl - EDDY Activation (Experimental): Following 2 mL irrigation with 5.25% NaOCl, EDDY activation was performed (as described in Arm 2), with 1 mL NaOCl used between activations. Final irrigation was performed with 2 mL saline and 2 mL 17% EDTA.
  Interventions: Device: EDDY Sonic Activation System
- 5.25% NaOCl - Passive Ultrasonic Irrigation (Experimental): After irrigation with 2 mL of 5.25% NaOCl, canals were activated using a passive ultrasonic tip (as in Arm 3), with 1 mL NaOCl used between activations. Final irrigation consisted of 2 mL saline and 2 mL 17% EDTA.
  Interventions: Device: Passive Ultrasonic Irrigation (PUI)

INTERVENTIONS:
Device: EDDY Sonic Activation System — EDDY is a sonic irrigation activation system operating at 6,000 Hz frequency with a flexible polyamide tip (25/04). In endodontic procedures, the EDDY tip is inserted 2 mm short of the working length into the root canal and activated for 20 seconds in three consecutive cycles. The sonic activation enhances irrigant agitation through cavitation and acoustic streaming, improving cleaning efficacy within the root canal system, especially in curved canals. The device does not contact dentin walls, reducing the risk of iatrogenic damage. In this study, EDDY was used to activate sodium hypochlorite solutions of either 2.5% or 5.25% concentration depending on the assigned group.
  Arms: 2.5% NaOCl - EDDY Activation; 5.25% NaOCl - EDDY Activation
Device: Passive Ultrasonic Irrigation (PUI) — Passive Ultrasonic Irrigation (PUI) involves the use of an ultrasonically activated file or tip inserted into the root canal 2 mm short of the working length, without contacting the dentinal walls. The ultrasonic tip is operated in a non-cutting, passive manner to generate acoustic streaming and cavitation within the irrigant. In this study, after initial irrigation with 2 mL of sodium hypochlorite (either 2.5% or 5.25%, depending on the group), ultrasonic activation was performed for 20 seconds in three consecutive cycles. Each activation was followed by 1 mL NaOCl irrigation. This method is designed to enhance the penetration and effectiveness of irrigants, especially in anatomically complex areas of the root canal system.
  Arms: 2.5% NaOCl - Passive Ultrasonic Irrigation; 5.25% NaOCl - Passive Ultrasonic Irrigation

SUMMARY:
The goal of this clinical trial was to evaluate the effect of different sodium hypochlorite (NaOCl) concentrations and irrigation activation techniques on the intensity of postoperative pain following single-visit root canal treatment in molar teeth with asymptomatic chronic apical periodontitis.

The primary research questions of this study were as follows:

Does using 2.5% or 5.25% sodium hypochlorite solution during root canal irrigation influence the severity of postoperative pain? Do activation techniques such as sonic activation using EDDY (a flexible polyamide tip-driven sonic irrigation device operating at 6,000 Hz; VDW GmbH, Munich, Germany) or passive ultrasonic irrigation (PUI) significantly reduce postoperative pain compared to conventional needle irrigation? In the non-activation groups, root canals were irrigated with 2.5% or 5.25% NaOCl using a 30-gauge side-vented needle without any further activation.

In the EDDY groups, root canals were irrigated using 2.5% or 5.25% NaOCl, followed by activation with a flexible polyamide EDDY tip (25/04) at 6,000 Hz, three times for 20 seconds.

In the PUI groups, root canals were irrigated using 2.5% or 5.25% NaOCl, and then subjected to passive ultrasonic activation with a suitable ultrasonic tip three times for 20 seconds, without contacting dentinal walls.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 16 and 60 years
* Systemically healthy individuals
* Presence of mandibular or maxillary first or second molar diagnosed with asymptomatic chronic apical periodontitis
* Negative response to electric pulp test, cold test, percussion and palpation tests
* Teeth eligible for single-visit root canal treatment
* Patients who provided written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding individuals
* Patients with uncontrolled systemic diseases (e.g., uncontrolled hypertension, uncontrolled diabetes mellitus, chronic renal failure, hematologic disorders)
* Patients undergoing chemotherapy or radiotherapy
* Individuals with infective endocarditis or immunosuppressive conditions
* Patients requiring antibiotic prophylaxis prior to dental treatment
* Use of anti-inflammatory or analgesic medications within 24 hours before treatment
* Teeth with calcified canals, internal/external resorption, or root fractures
* Patients unable to attend follow-up appointments or complete pain assessment forms

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | up to 72 hours
  The visual analog scale for pain is a straight line with one end meaning no pain (0) and the other end meaning the worst pain (10) imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine. Also called VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Koray Yılmaz, DDS MSc, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erkan E, Gundogar M, Uslu G, Ozyurek T. Postoperative pain after SWEEPS, PIPS, sonic and ultrasonic-assisted irrigation activation techniques: a randomized clinical trial. Odontology. 2022 Oct;110(4):786-794. doi: 10.1007/s10266-022-00700-0. Epub 2022 Mar 10. PMID 35267110